CLINICAL TRIAL: NCT02557191
Title: Biomarkers to Predict Neurodevelopmental Outcomes in Very Preterm Infants
Brief Title: Biomarkers, Neurodevelopment and Preterm Infants
Status: Terminated | Type: Observational
Why Stopped: Difficulty recruiting patients
Sponsor: Montefiore Medical Center (Other)
Collaborators: Albert Einstein College of Medicine (Other)
Responsible Party: Principal Investigator, Mamta Fuloria, Associate Professor, Pediatrics, Montefiore Medical Center
Other Study IDs: 2015-4484
Record Dates: First submitted 2015-07-06; First posted 2015-09-23 (Estimated); Last update posted 2019-04-25 (Actual); Status verified 2019-04

CONDITIONS: Preterm; Neurodevelopmental Disorder; Epigenetic Changes
MeSH Terms: conditions — Premature Birth; Neurodevelopmental Disorders | interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Biospecimen Retention: Samples With DNA — Cord blood, buccal swab and urine samples will be collected from enrolled patients.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Group 1: Preterm infants <32 weeks gestational age
  Interventions: Other: Observational study

INTERVENTIONS:
Other: Observational study

SUMMARY:
Approximately 2% of neonates in the US are born very preterm. Preterm births are associated with impaired cognitive, language and motor function, and increased risk for autism spectrum disorders. Epidemiological studies indicate a dose-response relationship between gestational age at delivery and cognitive impairments, with the most immature of newborns being the most susceptible to developmental delays. Sensitive and reproducible biomarkers of long-term neurocognitive impairments are currently lacking. The investigators seek to identify epigenetic markers that mediate the relationship between adverse prematurity-related exposures and neurocognitive impairments. The overarching hypothesis of this proposal is that DNA methylation profiles of CD34+ hematopoetic progenitor and stem cells from very preterm infants can be used as a risk-stratifying biomarker for predicting neurocognitive impairment in childhood.

ELIGIBILITY:
Inclusion Criteria:

* <32 weeks" gestation
* Born at Weiler Division of Montefiore

Exclusion Criteria:

* Intraventricular hemorrhage
* Chromosomal abnormalities
* Congenital viral conditions

Ages: 1 Day to 2 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Preterm infants <32 weeks GA
Sampling Method: Probability Sample
Enrollment: 4 (Actual)
Dates: Start 2015-04 (Actual); Primary Completion 2018-12 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Brain white matter development | 38-42 weeks adjusted age
  Brain MRI

SECONDARY OUTCOMES:
Neurodevelopment | 38-42 weeks adjusted age
  Administration of NICU Neonatal Neurobehavioral Scale
Neurodevelopment | 18-24 months adjusted age
  Administration of Bayley Scales of Infant and Toddler Development, 3rd edition

CONTACTS AND LOCATIONS:
Overall Officials: Mamta Fuloria, MD, Principal Investigator — Montefiore Medical Center
Locations (1):
- Jack D. Weiler Hospital, The Bronx, New York, United States